CLINICAL TRIAL: NCT03045224
Title: Endovascular Treatment in Patients With Peripheral Artery Disease: Real Life Effectiveness Off the Road of Studies PTA-Registry, a Prospective, Multicenter Study With 24-Month Follow-up
Brief Title: PTA-Registry, a Prospective, Multicenter Study With 24-Month Follow-up
Acronym: PTAReg
Status: Completed | Type: Observational
Sponsor: Vascular Center Berlin (Other)
Collaborators: BVMed - The German Medical Technology Association (Unknown); German Society for Angiology - Society for Vascular Medicine (DGA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. K.-L. Schulte, Head of Vascular Center Berlin, Vascular Center Berlin
Other Study IDs: 10PTAReg2016
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Efficacy/Long-term Effectiveness Endovascular Therapy in PAD
Keywords: PAD, PTA, mortality, morbidity, amputation rate, quality of life; Percutaneous transluminal angioplasty (PTA), Stenting, balloon angioplasty
MeSH Terms: conditions — Truncus Arteriosus, Persistent | interventions — Angioplasty, Balloon; Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PTA, balloon angioplasty, stent

SUMMARY:
The PTA-Registry (PTA-REG) is a prospective health services research registry to monitor and follow-up patients with peripheral arterial disease undergoing endovascular peripheral intervention. The PTA-REG has an interdisciplinary approach: cardiologists, angiologists, and radiologists contributed actively to this registry.

DETAILED DESCRIPTION:
The registry was created for the following purposes: evaluation of the clinical effectiveness, safety and quality of the endovascular therapy, and history of the disease after endovascular therapy. The resulting specific research questions were determination of the technical and clinical success of the procedure, monitoring of periinterventional complications, evaluation of vessel patency, amputation rate, mortality, and major adverse cardiac events during the follow-up. In addition, the quality of life after endovascular peripheral intervention over a period of two years was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* peripheral arterial disease of the iliac and lower extremity arteries and appropriate clinical indication for treatment with PTA according to current guidelines

Exclusion Criteria:

* no exclusion criteria and no age restriction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with peripheral arterial disease of the iliac and lower extremity arteries and appropriate clinical indication for treatment with PTA according to current guidelines were included in the registry. Presence of written informed consent for participating in the registry was mandatory. There were no exclusion criteria and no age restriction.
Sampling Method: Probability Sample
Enrollment: 1760 (Actual)
Dates: Start 2008-08; Primary Completion 2014-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
death of any cause | 2 years
revascularization (TLR, TVR) | 2 years

SECONDARY OUTCOMES:
minor or major amputation | 2 years
major adverse cardiac events and stroke | 2 years
quality of life | 2 years
  The follow-up was performed at months 6, 12, 18, and 24. The follow-up consisted of a quality of life questionnaire (EQ-5D)

IPD SHARING:
Plan to Share IPD: No